CLINICAL TRIAL: NCT06774157
Title: Evaluation of the Efficacy of the ALLYANE Procedure in the Treatment of Central Motor Inhibition Immediately After Knee Sprain as an Adjunct to Conventional Treatment.
Brief Title: Evaluation of the Efficacy of the ALLYANE Procedure in the Treatment of Central Motor Inhibition
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Allyane (Industry)
Collaborators: Orthopedic Center Santy, Lyon, France (Unknown); Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMI_LCA
Record Dates: First submitted 2024-10-07; First posted 2025-01-14 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Arthrogenic Muscle Inhibition; Arthrogenic Muscle Inhibitions
Keywords: AMI; ALLYANE; low frequency sounds; motor imagery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Management (Active Comparator): This group of patients will receive the conventional approach for managing motor inhibitions, which may include traditional physical therapy, exercises, and other rehabilitative techniques without any additional intervention.
  Interventions: Other: Standard management - Control group
- Standard Management + ALLYANE Process (Experimental): This group will receive the same standard management as the first group but with the addition of the ALLYANE process, a neuro-motor reprogramming technique designed to enhance muscle activation and re-establish motor control.
  Interventions: Other: A session combining motor imagery and listening to low frequency sounds; Other: Standard management - Control group

INTERVENTIONS:
Other: A session combining motor imagery and listening to low frequency sounds — Prospective study of the efficacy of the Allyane procedure after knee sprain
  Other Names: ALLYANE; Motor imagery; low frequency sounds
  Arms: Standard Management + ALLYANE Process
Other: Standard management - Control group — Active extension (e.g. by lateral raising of the quadriceps, strengthening of the quadriceps) quadriceps)
Other: Standard management - Control group — Flexor inhibition (e.g. massage, hamstring stretching)
Other: Standard management - Control group — Active flexion (e.g. strengthening the flexors)

SUMMARY:
The goal of this clinical study is to determine the effectiveness of restoring muscle strength in the management of motor inhibition when complemented by the ALLYANE process (neuro-motor reprogramming) compared to a standard management approach.

The main questions it aims to answer are:

* Does the ALLYANE process lead to greater muscle strength gains compared to standard care?
* Is there a functional benefit when standard management is complemented by the ALLYANE process?

The investigators will compare the group receiving standard care complemented by ALLYANE to a group receiving only standard care to evaluate if the ALLYANE process provides additional effects.

Participants will:

* Undergo assessments of muscle strength.
* Receive either standard management or standard management with ALLYANE.
* Complete functional evaluations before and after treatment.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of motor inhibition management using two different approaches: standard management alone and standard management supplemented by the ALLYANE neuro-motor reprogramming process. To ensure robust and reliable results, the study proposes enrolling a total of 120 patients, divided into two groups of 60 patients each.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 35 years
* No neurological history
* Have had a primary knee sprain
* Present with VMO lateralisation with or without the presence of flessum
* Quadricipital weakness between the healthy and injured limb of 50% or more as measured by a portable dynamometer
* Member of a social security scheme

Exclusion Criteria:

* Recurrent sprain
* Bilateral sprain
* Persons under guardianship, trusteeship or any other measure depriving them of their rights or liberty, and adults protected by law.
* Persons who do not understand French
* Knee trauma other than sprain
* Exclusion criteria for the Allyane procedure (COPHOSIS, cognitive difficulties, purely mechanical limitation)
* Algodystrophy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Muscle activity | Before and 3 weeks after conventional therapy
  Electromyography (EMG) during maximal voluntary isometric contraction of leg extension.

SECONDARY OUTCOMES:
Strength | Before and 3 weeks after conventional therapy
  Dynamometer during maximal voluntary isometric contraction of leg extension.

OTHER OUTCOMES:
Lysholm Questionnaire | Before and 3 weeks after conventional therapy.
  A self-administered survey used to evaluate knee function and stability.

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric Guillot, Pr, Study Chair — Laboratoire Interuniversitaire de Biologie de la Motricité
Locations (1):
- Centre Expert du Mouvement, Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
The shared IPD will include key data points such as demographic information, muscle strength assessment results, functional evaluation scores, and patient-reported outcomes like Lysholm Questionnaire results. Personal identifiers will be removed to ensure participant confidentiality. Data sharing will adhere to ethical and legal requirements. Specifically, the individual participant data sets underlying results in a publication will be shared.
Supporting Information: Study Protocol
Time Frame: The IPD and supporting information will be made available starting after statistical analysis is complete and during the process of writing the manuscript for publication. The data will remain accessible for a period of three years following the publication of the study results.
Access Criteria: Access to the IPD and supporting information will be granted to qualified researchers affiliated with academic, governmental, or non-profit institutions. They will have access to de-identified individual participant data, including demographic details, muscle strength assessments, functional evaluation results, and patient-reported outcomes. Access will be provided through a secure repository or data-sharing platform after approval of a data-sharing agreement. Researchers must agree to use the data solely for academic and non-commercial purposes, comply with all ethical guidelines, and acknowledge the source in any resulting publications.

REFERENCES:
- [Background] Dos Anjos T, Gabriel F, Vieira TD, Hopper GP, Sonnery-Cottet B. Neuromotor Treatment of Arthrogenic Muscle Inhibition After Knee Injury or Surgery. Sports Health. 2024 May-Jun;16(3):383-389. doi: 10.1177/19417381231169285. Epub 2023 Apr 27. PMID 37102673
- See also: Additional information about the ALLYANE method, which combines motor imagery and low-frequency sound, can be found on the website: http://allyane.com — http://allyane.com